CLINICAL TRIAL: NCT01664000
Title: A Phase 1, Open-Label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of Kevetrin (Thioureidobutyronitrile) Administered Intravenously, in Patients With Advanced Solid Tumors
Brief Title: A Safety, Pharmacokinetic and Pharmacodynamic Study of Kevetrin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellceutix Corporation (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTIX 12-101; 12-151 (Other: Dana-Farber Cancer Institute)
Record Dates: First submitted 2012-08-02; First posted 2012-08-14 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumors
Keywords: Tumors; carcinoma; apoptosis; p53; p21; Caspase3; PARP; MDM2; PUMA
MeSH Terms: conditions — Neoplasms; Carcinoma; Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kevetrin (Experimental): thioureidobutyronitrile intravenous once/week for 3 weeks/ cycle
  Interventions: Drug: thioureidobutyronitrile

INTERVENTIONS:
Drug: thioureidobutyronitrile — Kevetrin (thioureidobutyronitrile)
  Other Names: Kevetrin

SUMMARY:
In the laboratory, Kevetrin activates p53, a tumor suppressor protein that has an important role in protecting the body. p53 functions by activating proteins that repair DNA and kill cells that have genetic mutations such as in cancers. Research experiments showed that when cancer cells were treated with Kevetrin, it activated p53 which induced p21, a protein that inhibits cancer cell growth. p53 also induced PUMA (p53 up-regulated modulator of apoptosis), a protein that causes tumor cell death. Because of these activities, slowing cancer cell growth and causing cancer cell death, Kevetrin may help to treat tumors.

DETAILED DESCRIPTION:
Kevetrin was found to be effective in pre-clinical studies of human xenograft tumor models and was reasonably well-tolerated at therapeutic doses in the non-clinical animal studies. Kevetrin was also effective in multi-drug resistant tumor models; therefore, Kevetrin has the potential to treat tumors that have become resistant to standard chemotherapy. This trial will determine tolerance in humans and, possibly, efficacy with a Phase I, open-label, dose-escalation, safety, pharmacokinetic, and pharmacodynamic study of Kevetrin, in adult patients with solid tumors.

The primary objectives are the following:

* To determine the maximum tolerated dose (MTD) of Kevetrin.
* To determine the dose limiting toxicities (DLT) of Kevetrin.
* To establish a safe dose level of Kevetrin that can be used for future studies.

The secondary objectives are to determine the following:

* The pharmacokinetics of Kevetrin in humans.
* Observe for evidence of antitumor activity following administration of Kevetrin.
* If Kevetrin induces changes in the biomarker p21 in peripheral blood lymphocytes.
* If there is a pharmacodynamic relationship between the plasma concentrations of Kevetrin and a clinical or cellular effect.

During each 4 week cycle, each patient will receive three weekly doses of Kevetrin given as a 1 hour intravenous infusion followed by a 1 week off-treatment period. Following each dose, each patient will be monitored. If the patients have acceptable safety and tolerance, Kevetrin will be given once weekly for a total of 3 weeks. During each cycle patients will be evaluated for safety, tolerance, and Dose-Limiting Toxicity (DLT) that occur during a cycle.

ELIGIBILITY:
Inclusion Criteria:

* Males / females, ≥ 18 years old, any race / ethnicity, who can provide written Informed Consent
* Life expectancy ≥ 3 months
* Pathologically confirmed solid tumor, locally advanced / metastatic, refractory after standard therapy, or for which no effective curative or surgical treatment options are available
* Measurable disease on baseline imaging per RECIST 1.1 criteria
* ECOG performance status ≤ 1
* Liver function:
* Bilirubin ≤ 1.5 X upper limit of normal
* AST, SGOT, ALT, SGPT ≤ 2.5 X upper limit of normal, < 5 upper limit if there are liver metastases
* Renal function:
* Serum creatinine within normal limits
* Hematologic status:
* Absolute neutrophil count ≥ 1500 cells/mm3.
* Platelet count ≥ 100,000/mm3.
* Hemoglobin ≥ 9 g/dL
* Coagulation status:
* Coagulation Prothrombin time ≤ 1.5 X upper limit
* Partial thromboplastin time ≤ 1.5 X upper limit
* Males must agree to use condoms during sex to prevent spillage of semen for the duration of the study and for 3 months after the patient leaves the study
* Females in the study must not be pregnant or breast feeding and not planning to become pregnant or breast feed for the duration of the study, and for at least three months after study completion
* Women of childbearing potential must commit to using a double barrier method of contraception, an intrauterine device, or sexual abstinence for the duration of the study and for at least three months after study completion
* Serum pregnancy test for women of child bearing potential must be negative at entry into study
* Written voluntary informed consent: the patient is capable of complying with the requirements of the written Informed Consent Form and complying with protocol requirements

Exclusion Criteria:

* History of significant disease that in the Investigator's opinion would put the patient at high risk on the trial
* Cognitive impairment sufficient to render the patient incapable of giving informed consent
* History of clinically significant psychiatric illness that would prevent the patient from providing a valid ICF and complying with protocol requirements
* Unwillingness or inability to comply with procedures required in this protocol
* History or presence of alcoholism or drug abuse within the past 2 years
* Patients who have had a major surgical procedure within the past 6 weeks
* History of HIV, hepatitis B, or hepatitis C
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy
* Women of childbearing potential who are lactating, pregnant or there is the likelihood of becoming pregnant within the coming 12 months; a positive serum beta-human chorionic gonadotropin test at time of screening for entry into study
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Patients with a mean QTc interval greater than 480ms are excluded. Avoid concomitant administration of agents that prolong the QT interval, except at the discretion of the investigator. If advised, patients should discontinue the use of these agents at least 2 weeks before the study begins. No uncontrolled arrhythmias.
* Patients currently receiving other investigational agents
* Participation in a study of an investigational drug within 4 weeks prior to the planned first day of study drug administration
* Patients who have undergone radiation within the past 4 weeks
* Treatment with molecularly targeted agents within the past 3 weeks prior to planned first study drug administration. Patients who were receiving standard chemotherapy or experimental therapies must wait 4 weeks from their last dose prior to the planned first study drug administration. Patients treated with nitrosoureas or mitomycin C must wait 6 weeks from their last dose prior to the planned first study drug administration.
* Patients with known brain metastases may be excluded from this study. However, patients may be eligible if scans show limited disease or repeat scans show stable disease in the opinion of the investigator and patients have no ill effect from the metastases.
* Herbal supplements are prohibited 1 week prior to the planned first study drug administration, during the clinical study, and up to the time that the patient is discharged from the study
* Patients who have been exposed to medications, herbal preparations, or foods known to be predominant Cytochrome P450 2C9, 2C19, 2D6, 3A4/5 substrates, strong inhibitors or inducers within 7 days of planned first study treatment day
* Patients who in the opinion of the Investigator would not be able to provide reliable study data or be available for study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Kevetrin | up to 6 months
  A dose will be declared the MTD if at least 1 patient out of 6 patients experience a dose limiting toxicity (DLT) at the highest dose level below the maximally administered dose. Once an MTD has been established, up to 12 additional patients may be enrolled at the MTD dose level for confirmation of safety.
  The maximally administered dose is if 1 or more of 6 patients experience a DLT.
Dose Limiting Toxicities (DLT) of Kevetrin. | up to 4 weeks
  The definition of dose limiting toxicity (DLT) is in accord with the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE). Dose limiting toxicity will be defined as:
  * Grade 3 or 4 neutropenia complicated by fever, or greater than 38.5°C documented infection, or Grade 4 neutropenia of greater than 7 days duration
  * Grade 4 thrombocytopenia or grade 3 thrombocytopenia complicated by hemorrhage
  * Any grade greater than 3 non-hematologic toxicity unless there is clear alternative evidence that the adverse event (AE) was not caused by Kevetrin
  * Grade 3 diarrhea, nausea, or vomiting may be excluded from dose-limiting toxicities provided that the maximum time limit for supportive measures is 48 hours.

SECONDARY OUTCOMES:
Pharmacokinetic Profile of Kevetrin | Day 1 Pre-dose, 30 minutes after starting the infusion, 1 hr, 1 hr 10 min, 1 hr 20 min, 1 hr 30 min, 1 hr 45 min, 2 hr, 2 hr 30 min, 3 hr, 4 hr, 5 hr, 7 hr, and 24 hr after the initiation of the infusion
  The pharmacokinetics (PK) of Kevetrin will be determined for all patients enrolled in the study on Day 1 of Cycle 1 and Day 15 of Cycle 2. Blood samples will be obtained before dosing, 30 minutes after starting the infusion, 1 hr, 1 hr 10 min, 1 hr 20 min, 1 hr 30 min, 1 hr 45 min, 2 hr, 2 hr 30 min, 3 hr, 4 hr, 5 hr, 7 hr, and 24 hr after the initiation of the infusion.
  The pharmacokinetic profile will be analyzed by standard noncompartmental methods to provide estimated values of the pharmacokinetic parameters and associated variables, such as area under the plasma concentration versus time curve (AUC) and peak plasma concentration (Cmax) of Kevetrin. Associations between pharmacokinetic variables and drug-related toxicities will be evaluated.
Pharmacokinetic Profile of Kevetrin | Day 15 Pre-dose, 30 minutes after starting the infusion, 1 hr, 1 hr 10 min, 1 hr 20 min, 1 hr 30 min, 1 hr 45 min, 2 hr, 2 hr 30 min, 3 hr, 4 hr, 5 hr, 7 hr, and 24 hr after the initiation of the infusion
  The pharmacokinetics (PK) of Kevetrin will be determined for all patients enrolled in the study on Day 1 of Cycle 1 and Day 15 of Cycle 2. Blood samples will be obtained before dosing, 30 minutes after starting the infusion, 1 hr, 1 hr 10 min, 1 hr 20 min, 1 hr 30 min, 1 hr 45 min, 2 hr, 2 hr 30 min, 3 hr, 4 hr, 5 hr, 7 hr, and 24 hr after the initiation of the infusion.
  The pharmacokinetic profile will be analyzed by standard noncompartmental methods to provide estimated values of the pharmacokinetic parameters and associated variables, including area under the plasma concentration versus time curve (AUC) and peak plasma concentration (Cmax) of Kevetrin. Associations between pharmacokinetic variables and drug-related toxicities will be evaluated.
Change in tumor size | baseline and 2 months
  Change in tumor size based on RECIST criteria version 1.1. using MRI, CT scan, and/or standard of care imaging
Change in tumor size | baseline and 4 months
  Change in tumor size based on RECIST criteria version 1.1. using MRI, CT scan, and/or standard of care imaging
Change in tumor size | baseline and 6 months
  Change in tumor size based on RECIST criteria version 1.1. using MRI, CT scan, and/or standard of care imaging
Decrease in serum tumor marker | baseline and 1 month
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Decrease in serum tumor marker | baseline and 2 months
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Decrease in serum tumor marker | baseline and 3 months
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Decrease in serum tumor marker | baseline and 4 months
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Decrease in serum tumor marker | baseline and 5 months
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Decrease in serum tumor marker | baseline and 6 months
  A decrease in a tumor marker in the serum may also suggest evidence of anti-tumor efficacy. The following tumor markers will be evaluated: Carcinoembryonic antigen (CEA), Cancer Antigen 125 (CA125), Cancer Antigen 19-9 (CA19-9), Cancer Antigen 15-3 (CA15-3), Prostate Specific Antigen (PSA), or other appropriate markers. The choice of the individual tumor markers will be based on the type of tumor of the patient and the testing that has preceded the patient's participation in this study.
Changes in the biomarker p21 in peripheral blood lymphocytes | baseline and 7 hours
  For biomarker analysis, p21 expression, assayed by qPCR, in peripheral blood lymphocytes after Kevetrin administration.
Changes in the biomarker p21 in peripheral blood lymphocytes | baseline and 24 hours
  For biomarker analysis, p21 expression, assayed by qPCR, in peripheral blood lymphocytes after Kevetrin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber / Beth Israel Deaconess Medical Center / Harvard Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes